CLINICAL TRIAL: NCT01064726
Title: A Double Blind (3rd Party Open), 3-Way Crossover Study To Explore The Reproducibility Of Inflammatory Markers After Nasal Allergen Challenge In Subjects With Seasonal Allergic Rhinitis (Out Of Season) And The Effect Of A Single Dose Of Ibuprofen Or Fluticasone Propionate On The Allergen Response.
Brief Title: A Study To Explore The Effect On Inflammatory Markers After Nasal Allergen Challenge In Subjects With Seasonal Allergic Rhinitis And The Effect Of A Single Dose Of Ibuprofen Or Fluticasone Propionate On The Allergen Response.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A9011065
Record Dates: First submitted 2009-09-21; First posted 2010-02-08 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-06

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis Nasal Allergen Challenge Inflammatory Markers
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Ibuprofen; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ibuprofen (Experimental)
  Interventions: Drug: Ibuprofen
- Fluticasone propionate (Experimental)
  Interventions: Drug: Fluticasone propionate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen — 800 mg oral
  Arms: Ibuprofen
Drug: Fluticasone propionate — 200 mcg intra-nasal
  Arms: Fluticasone propionate
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
After a nasal allergen challenge it should be possible to measure markers of inflammation that may be useful to assess the properties of future drugs. If these markers are reproducible and impacted by the study drugs they could be useful for future drug development.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with seasonal allergic rhinitis (out of season).
* Sensitive to ragweed skin prick test and screening nasal allergen challenge.

Exclusion Criteria:

* Subjects with significant concomitant diseases.
* Subjects with symptoms of allergic rhinitis in 2 weeks prior to screening.
* Female subjects that are pregnant or nursing. Subjects with hypersensitivity to study drugs or allergen challenge.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Nasal inflammatory markers | 8h 45 min post dose
Acoustic rhinometry | 8h 45 min post dose
Nasal symptom scores | 8h 45 min post dose

SECONDARY OUTCOMES:
Spirometry | 8h 45 min post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Omaha, Nebraska, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9011065&StudyName=A%20Study%20To%20Explore%20The%20Effect%20On%20Inflammatory%20Markers%20After%20Nasal%20Allergen%20Challenge%20In%20Subjects%20With%20Seasonal%20Allergic%20Rhinitis%20And%20T